CLINICAL TRIAL: NCT02970279
Title: Effect of Treatment Augmentations Embedded in Behavioural Activation Group Therapy on Reducing Drop-out and Stasis Rates in Depression
Brief Title: Reducing Stasis Outcomes for Depression in Group Behavioural Activation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Collaborators: Sheffield Health and Social Care NHS Foundation Trust (Unknown); Howard Morton Trust (Unknown)
Responsible Party: Principal Investigator, Melanie Simmonds-Buckley, PhD Research Student, University of Sheffield
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol Version 3.0
Record Dates: First submitted 2016-11-11; First posted 2016-11-21 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Depression
Keywords: Behavioural activation; Psychotherapy, group; Depression; Depressive disorder
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enhanced Behavioural Activation Groups (Experimental): Behavioural activation group (BAG) psychotherapy delivered with two embedded treatment augmentations;
  1. Implementation intentions
  2. Dose-response psychoeducation
  Interventions: Behavioral: Behavioural Activation Group (BAG) Psychotherapy

INTERVENTIONS:
Behavioral: Behavioural Activation Group (BAG) Psychotherapy — Behavioural activation (BA) is a psychotherapy intervention based on behaviour theory and operant conditioning. It teaches patients to reduce avoidant depressive behaviours and in turn increase the positive reinforcement they receive from their environment for non-depressive behaviours through the use of activity scheduling and pleasant events. For the trial, BA will be delivered in a group format (BAG) and facilitated by two therapists. BAG treatment will consist of eight weekly sessions, lasting two hours and will follow a manualised treatment protocol. Each session will be based on a different topic relevant to the principles of BA and patients will be given between session work to complete to encourage increased participation in rewarding personally meaningful activities.

SUMMARY:
Depression is one of the most common mental health disorders and it is estimated up to 50% of patients do not respond to evidenced-based psychotherapy treatment, recording a 'stasis' outcome. However, there is limited research understanding this population, meaning a considerable number of people continue to suffer. The purpose of this study is to 1) identify depression stasis prevalence and predictors in an existing evidenced-based group treatment for depression, 2) run a clinical trial to test whether an embedded intervention based on theoretical and clinical practice evidence can help reduce patient depression stasis and drop-out rates and 3) understand what aspect of therapy produces change (or prevents change in stasis). The study will be based on behavioural activation (BA) therapy delivered in an eight-session group format in an Improving Access to Psychological Therapies (IAPT) service in the United Kingdom. BA is one of the most effective psychotherapies available for depression and focuses on helping patients to increase their engagement with valued activities to help break out of the cycle of depression. Firstly, an archived anonymised dataset of routine depression measures from patients who have previously received the existing group BA treatment will be analysed. Secondly, the group BA treatment delivered to patients in 2017 will be enhanced with two treatment augmentations. One augmentation will target stasis outcomes through the addition of specific 'if-then' planning (known as implementation intentions) when setting between-session homework and the other augmentation will target patient drop-out by informing patients about group BA effectiveness and therapy-dose evidence. The stasis outcomes and drop-out rates from the enhanced treatment in the trial will be compared with the archived outcomes to see if the intervention has had an effect and the role of engaging in valued living as a mechanism of change for depression symptoms will be examined. It is hypothesised that a) 50% of patients who have received the existing BA group treatment for depression will have a stasis outcome, b) there will be a significant reduction in depression stasis outcomes and drop-out rate following the enhanced BA group treatment delivered in the trial and c) engagement in valued living will have a mediating effect on outcome for responding patients following the enhanced BA group treatment but the effect will not be present for patients with a stasis outcome.

DETAILED DESCRIPTION:
A one-armed quasi-experimental trial will be used to test the effect of two embedded behavioural activation group (BAG) treatment augmentations on treatment outcomes and to identify a potential outcome mediator for patients with a stasis outcome. A non-randomised design enables data to be collected which reflects routine clinical practice and address stasis outcomes as they occur in real-world services. A matched pairs design will be implemented in the analysis to allow comparison of the enhanced BAG data with historical control data from archived outcomes of the existing treatment (i.e. the baseline data).

Patients who access the Improving Access to Psychological Therapies (IAPT) service in Sheffield, United Kingdom with a primary presenting problem of depression and are referred to BAG will be approached to take part in the study. Patients will be asked to provide informed consent to agree for their weekly routine outcome scores from enhanced BAG to be used in the study.

Enhanced BAG Augmentations

The existing BAG treatment will be enhanced with embedded treatment augmentations. The augmentations will consist of two strands; 1) implementation intentions to directly target reducing stasis and 2) psychoeducation to target reducing drop-out.

Implementation Intentions: The first augmentation will be a top-down theoretically informed 'implementation intentions' enhancement to target reducing the stasis outcome rate. Implementation intentions are specific plans about how, when and where goals will be acted upon, formed using an if-then format in order to effectively implement actions. Patients will be taught to use if-then planning (implementation intentions) to help them complete the between-session which is crucial to producing change in BA.

Dose-Response Psychoeducation: The second augmentation will be a dose-response psychoeducation enhancement aimed at reducing the dropout rate. Patients will be given information based on practice-based evidence about the effectiveness of BAG and dose-response information (minimum number of sessions required to experience change).

Treatment Integrity

Treatment adherence to the protocol will be assessed using a BAG adherence checklist created for this trial. Adherence will be checked and compared using self-report and an expert rater; i) after each session the BAG facilitators will complete the session integrity measure to check self-report adherence and ii) the BAG facilitator lead will observe and rate one session from each course of BAG to provide an expert adherence check.

Data Collection

Data collection for the study will run for a year from January 2017 until December 2017 incorporating six BAG treatment groups.

Data Analysis

The data will be analysed using the intention-to-treat (ITT) principle. The final available measure will be used as the post score or if there is only one score available, it will be assumed there was no change. Patients who do not score above the clinical cut-off for depression (score of ≥10 on Patient Health Questionnaire [PHQ-9]) prior to commencing BAG will not be included in the analysis to avoid a floor effect when calculating stasis outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who access the Sheffield Improving Access to Psychological Therapies (IAPT) service (United Kingdom) with depression as the primary presenting problem
* Patients with co-morbid anxiety symptoms can be included as long as depression is the primary diagnosis
* Are referred to and choose the Behavioural Activation Group (BAG) treatment option
* Able to attend the BAG intervention
* Aged 18 or over

Exclusion Criteria:

* Primary diagnosis that is not depression
* Patients who do not choose BAG as a treatment option
* Aged under 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9) scores | Week 1 (pre-treatment), at every weekly treatment session attended (for 8 weeks) and at week 8 (end of treatment)
  Validated 9-item self-report measure of depressive symptoms

SECONDARY OUTCOMES:
Patient attendance at treatment sessions | Weeks 1-8 (every weekly treatment session - maximum of 8)
  Number of therapy sessions patients attend in a course of treatment
Change in Valued Living Questionnaire (VLQ) score | Week 1 (pre-treatment), week 4 (at the 4th treatment session) and at week 8 (end of treatment)
  Validated self-report measure of engagement in valued living
Change in Generalised Anxiety Disorder Assessment (GAD-7) score | Week 1 (pre-treatment), at every weekly treatment session attended (for 8 weeks) and at week 8 (end of treatment)
  Validated 7-item self-report measure of anxiety symptoms
Change in Work and Social Adjustment Scale (WSAS) score | Week 1 (pre-treatment), at every weekly treatment session attended (for 8 weeks) and at week 8 (end of treatment)
  Validated self-report measure of functional impairment as a result of mental health problems

OTHER OUTCOMES:
Behavioural activation group (BAG) therapy adherence | Weeks 1-8 (Every treatment session)
  BAG facilitators will complete an therapy adherence checklist (designed for this trial) after each session. An external rater will rate one session of each course of treatment to ensure adherence to the treatment protocol

CONTACTS AND LOCATIONS:
Overall Officials: Melanie K Simmonds-Buckley, BSc, Principal Investigator — University of Sheffield; Stephen Kellett, DClinPsy, Principal Investigator — University of Sheffield & Sheffield Health and Social Care NHS Foundation Trust; Glenn Waller, PhD, Principal Investigator — University of Sheffield
Locations (1):
- Sheffield Health and Social Care NHS Foundation Trust - Improving Access to Psychological Therapies Service, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The data will be anonymised and analysed collectively so individual participant data will not be identifiable within any reports or publications.

REFERENCES:
- [Background] Gollwitzer, P. M. (1999). Implementation intentions: Strong effects of simple plans. American Psychologist, 54, 493-503.